CLINICAL TRIAL: NCT05200702
Title: Assessment of Safety and Acute Effects of a Knee-hip Powered Soft Exoskeleton in Patients With Neuromuscular Disorders
Acronym: Exo-NMD1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Exo-NMD1
Record Dates: First submitted 2021-12-02; First posted 2022-01-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Muscular Dystrophies; Congenital Myopathy; Idiopathic Inflammatory Myopathies; Mitochondrial Myopathies; Glycogen Storage Disease
Keywords: Neuromuscular disorders; Myopathy; Muscle; Exoskeleton; Device; Motion assistance; FSHD; LGMD
MeSH Terms: conditions — Muscular Dystrophies; Myotonia Congenita; Myositis; Mitochondrial Myopathies; Glycogen Storage Disease; Neuromuscular Diseases; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: Comparison of the results obtained during different standardized physical evaluations by patients and healthy subjects, with or without a movement assistance device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee-hip Powered Soft Exoskeleton (Experimental): Patients and healthy subjects will use a Knee-hip Powered Soft Exoskeleton to perform different standardised tasks
  Interventions: Device: Knee-hip Powered Soft Exoskeleton (MyoSuit, MyoSwiss, Zurich, Switzerland)
- No assistance device (No Intervention): Patients and healthy subjects will perform different standardised tasks without Knee-hip Powered Soft Exoskeleton

INTERVENTIONS:
Device: Knee-hip Powered Soft Exoskeleton (MyoSuit, MyoSwiss, Zurich, Switzerland) — Patients and healthy subjects will wear the movement assistance device to perform different standardised physical evaluations.
  Arms: Knee-hip Powered Soft Exoskeleton

SUMMARY:
The aims of the current study are as follow:

i) Evaluate the safety, usability, and acute efficiency of a powered knee-hip dermoskeleton (MyoSuit, MyoSwiss, Zurich, Switzerland) in patients with neuromuscular disorders, ii) Elaborate recommendations regarding usability criteria for safe and efficient use the device in patients with neuromuscular disorders (e.g. type and severity of patient's functional deficits), iii) generate necessary data to foresee a future study involving a home use of the device and assessment of long-term benefits.

DETAILED DESCRIPTION:
Patients with neuromuscular disorders display different type of symptoms depending on the type of pathology. Diseases like facioscapulohumeral dystrophy (FSHD), limb-girdle muscular dystrophy (LGMD2b), sporadic inclusion body myositis (SIBM) or Pompe disease (PD) are characterized by severe muscle weakness leading to reduced functional capacities. This leads to a dramatic decrease of quality of life (e.g. reduced autonomy/participation, social isolation, depression) associated with increased fall risk and complications (e.g. trauma, cardio-vascular issues, trauma, chronic pain, loss of bone mass, and weight gain).

However, a residual of level of strength and residual function may be maintained over years, even at severe disease stages allowing transfers and ambulation. However, the maintenance of this type of activity is often associated with substantial compensatory movements, leading to high load on joints, orthopedic complications, and high fall-risk.

In contrast to traditional passive assistive devices such as orthoses, powered assistive devices, frequently termed dermo- or exoskeletons, have a very high potential for compensating muscle weakness and regain mobility and independence. Devices such as the ReWalk or the Indego use rigid structures, in parallel to the user's legs, and electric motors to stabilize the human against gravity during standing and walking. Thus far, these systems have been used mostly in clinical environments for gait rehabilitation in neurological conditions (e.g. spinal cord injury, post-stroke syndrome). Their weight, which can range from 13 to 48 kg , can make them difficult to use and transport, thus limiting their applicability beyond clinical environments. However, for assistive devices to be used in everyday life, they must provide assistance across activities of daily living (ADLs) in an unobtrusive manner.

Wearable motion assistance systems, especially those dedicated to lower limbs are highly promising for ambulant patients with neuromuscular disorders (e.g. FSHD, LGMD, SIBM or PD). In these conditions, the prevalence of lower-limb muscle weakness, in particular in proximal muscle groups (i.e. providing strength/torque to hips and knees) is very high. Schmidt et al. recently introduced a powered knee-hip soft exoskeleton (the Myosuit), a soft, wearable device designed to provide continuous assistance at the hip and knee joint when working with and against gravity in ADLs. This robotic device combines active and passive elements with a closed-loop force controller designed to behave like an external muscle (exomuscle) and deliver gravity compensation to the user. With 5.6 kg including batteries, the Myosuit is one of the lightest untethered devices capable of delivering gravity support to the user's knee and hip joints. In healthy subject, the Myosuit has been shown to effectively assist its users in gravity-intensive ADLs, such as sitting transfers. However, the effect of the device on movement parameters and user perception must be clarified. We believe that ambulant patients with neuromuscular disorders can highly benefit from a system that provides mobility assistance like the Myosuit. The use of such a device has the potential to shift the loss of ambulation/transfer abilities to a higher age and might mitigate disease progression and occurrence of complications. Whether the Myosuit may be safe, usable, and efficient in ambulant patients with neuromuscular disorders, remain to be specifically investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and < 70 years of age
* Height between 1.50 m and 1.95 m
* Weight between 45 kg and 110 kg
* Abdominal perimeter < 125 cm
* Written informed consent
* Affiliate or beneficiary of a social security scheme
* Able to comply with all protocol requirements
* Confirmed diagnosis of a pathology belonging to one of the following family*:

  * Primary disorders of muscles

    * Muscular dystrophy
    * Congenital myopathies
    * Idiopathic inflammatory myopathy
    * Mitochondrial myopathies
  * Metabolic disorders

    * Inborn errors of metabolism
* Glycogen storage disease
* Functional capacities:

  * Able to stand up from a chair with armrest without other supports at least 3 times and at most 15 times in 30 seconds.
  * Report the ability to walk without the assistance of a person at least 2min
  * The use of traditional orthoses and walking aids will be accepted excepted knee orthoses and walkers (e.g. canes/crutches, ankle foot orthosis).

Exclusion Criteria:

* Unable to participate in the study
* Inability to comply with protocol requirements
* Guardianship/trusteeship
* Pregnant or nursing women
* Unstable Cardiomyopathy
* Symptomatic orthostatic hypotension
* Medical history of osteoporotic fracture
* Balance disorder with extra neuromuscular causes
* Recent trauma (fall, accident, ...)
* Unstable Cardiomyopathy
* Severe respiratory insufficiency
* Flexion contracture in the knee and hip joint in excess of 10°
* Varus malposition in excess of 10° or valgus malposition in excess of 10°

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Absence of adverse effect attributable to the use of the device during task performed within a knee-hip powered soft exoskeleton | Through study completion, on average 4 weeks

SECONDARY OUTCOMES:
Variation in the 2 Minutes Walking Test distance (express in meters) when performed using versus not using the device | Visit 2 and 3, on average 2 weeks
Variation in the 10 Meters Walking Test performance (express in seconds) when performed using versus not using the device | Visit 2 and 3, on average 2 weeks
Difference of performance with and without the device during 30 Sit To Stand | Visit 2 and 3, on average 2 weeks
Difference of performance with and without the device during simple Sit To Stand | Visit 2 and 3, on average 2 weeks
Difference of performance with and without the device during the squating test | Visit 2 and 3, on average 2 weeks
Difference of performance with and without the device during Time Up & Go test | Visit 2 and 3, on average 2 weeks
Difference of performance with and without the device during stairs climbing test | Visit 2 and 3, on average 2 weeks
Variation in spatiotemporal gait parameters during the 2 Minutes Walking Test with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Spatiotemporal gait parameters: Cadence, Gait Speed, Step Duration, Stride Length, Cadence Asymmetry, Gait Speed Asymmetry, Stance Asymmetry, Stride Length Asymmetry
Variation in spatiotemporal gait parameters during the 10 Meters Walking Test with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Spatiotemporal gait parameters: Cadence, Gait Speed, Step Duration, Stride Length, Cadence Asymmetry, Gait Speed Asymmetry, Stance Asymmetry, Stride Length Asymmetry
Variation in kinematics parameters during 30 Sit To Stand with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Kinematics parameters: Gait Joint Angles, Stick Plot Visualization - Sagital plane, Hip-Knee & Knee-Ankle Plots
Variation in kinematics parameters during unique Sit To Stand with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Kinematics parameters: Gait Joint Angles, Stick Plot Visualization - Sagital plane, Hip-Knee & Knee-Ankle Plots
Variation in kinematics parameters during Time Up & Go evaluation with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Kinematics parameters: Gait Joint Angles, Stick Plot Visualization - Sagital plane, Hip-Knee & Knee-Ankle Plots
Variation in kinematics parameters during stairs climbing test with and without the device using 3D accelerometers' system | Visit 2 and 3, on average 2 weeks
  Kinematics parameters: Gait Joint Angles, Stick Plot Visualization - Sagital plane, Hip-Knee & Knee-Ankle Plots
Modification of lower limb muscle recruitment measured by surface EMG with and without the device | Visit 2 and 3, on average 2 weeks
Variation in postural stability measured by force platform with and without the device | Visit 2 and 3, on average 2 weeks
  Mean Velocity, RMS Sway
Modification in scoring of the device measured by the Modified Nordic Questionnaire | Through study completion, on average 4 weeks
Positive scoring of device efficiency measured by the System usability scale | Through study completion, on average 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Myology, Paris, France

IPD SHARING:
Plan to Share IPD: No